CLINICAL TRIAL: NCT05546164
Title: Strength and Dexterity of Less Affected Hand of Hemiparetic Cerebral Palsy Children: A Comparison Study With Normal Peers
Brief Title: Strength and Dexterity of Less Affected Hand of Hemiparetic Cerebral Palsy Children
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mohamed Hassan, Principal Investigator, Cairo University
Other Study IDs: No: p.T. R E C /012 /003789
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Unilateral cerebral palsy; grip strength; pinch strength; upper limb dexterity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemiparetic group: This group will contains 60 children with hemiparesis
  Interventions: Other: Assessment of hand grip strength; Other: Assessment of pinch strength; Other: Assessment of upper limb dexterity
- Normal group: This group will contains 60 children with normal children
  Interventions: Other: Assessment of hand grip strength; Other: Assessment of pinch strength; Other: Assessment of upper limb dexterity

INTERVENTIONS:
Other: Assessment of hand grip strength — Assessment of hand grip strength
Other: Assessment of pinch strength — Assessment of pinch strength
Other: Assessment of upper limb dexterity — Assessment of upper limb dexterity

SUMMARY:
The contralateral hand deficits are often masked by the complex clinical presentation of the more affected hand in children with spastic hemiparesis. Thus, intervention targeting the contralateral hand is not often a component of the child's rehabilitation plan of care. The presence of bilateral hand deficits, even if subtle in the contralateral hand, may limit the transfer of unimanual gains following rehabilitation to bimanual activities of daily living tasks. However, conservation of upper-limb function of the less-affected side is highly important for individuals with hemiparesis, because this side is often employed as a compensatory 'tool' in performing activities of daily living . Therefore, the current study will be conducted to determine and compare the motor abilities of the less affected hand of children with hemiparesis.

DETAILED DESCRIPTION:
An impairment of the less affected hand of hemiparetic cerebral palsy children can be detrimental to the development of bimanual skills. It would be beneficial to identify and quantify the severity of any impairment of the less affected hand of hemiparetic cerebral palsy children. Hemiparetic cerebral palsy may present with substantial deficits in hand function, because bimanual activities involve the ability to use the affected and contralateral hands together for grasp and stabilization. Several authors have evaluated bimanual involvement in cerebral palsy but these studies have not compared the contralateral hand with norms. The less affected hand is widely regarded as "normal" or "unaffected" and is consequently rarely evaluated.

Several authors have reported incidental findings of subtle deficits in the less affected extremity, noted that hemiparetic children "also presented motor impairments in their non-paretic hand, especially in dexterity.

The purpose of this study is to assess the grip ,pinch strength and dexterity of less affected hand of hemiparetic cerebral palsy children and compare with dominant hand of normal peers

ELIGIBILITY:
Inclusion Criteria:

* Children will be recruited according to the following criteria:
* Age range between 6 and 10 years.
* Both sexes
* The degree of spasticity rang from grade 1 to 1+ according to Modified Ashworth scale (Appendix II).
* They can follow the order during the testing.

Exclusion Criteria:Children will be excluded from the study if they had any of the following criteria;

* Significant visual or auditory defect that may affect their performance.
* Previous orthopedic surgery for upper extremity.
* Injection with Botulinium toxin in the last 6 months.
* Structural deformities in any joint or bone of the upper limbs.
* Practicing any form of sports.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will include 120 children of both gender with age from 6 years to 10 years
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | from October 2022 to September 2023
  Hand dynamometer will be used to measure grip strength. It is a reliable tool, by measuring the amount of pressure applied to the compressible bulb-shaped rubber handle (Innes, 1999).The child sit in chair with armrest, suitable back support, feet flat on the floor, shoulder adducted to side, elbow flexed to 90 degree and forearm in neutral position then teach the child how to apply pressure on bulb through grip or pinch pressure for 3 times and their mean was calculated.
Hand pinch strength | from October 2022 to September 2023
  Hand dynamometer will be used to measure pinch strength. It is a reliable tool, by measuring the amount of pressure applied to the compressible bulb-shaped rubber handle (Innes, 1999).The child sit in chair with armrest, suitable back support, feet flat on the floor, shoulder adducted to side, elbow flexed to 90 degree and forearm in neutral position then teach the child how to apply pressure on bulb through grip or pinch pressure for 3 times and their mean was calculated.
upper limb dexterity | from October 2022 to September 2023
  Functional dexterity test will be used for assessment of fine motor dexterity. it is a timed pegboard test that provides objective assessment of in-hand manipulation and tripod pinch, .It consists of 16 cylindrical pegs arranged on a peg board in 4 rows of 4 pegs. Participants are instructed to pick up each peg, turn it over in their hand while refraining from supinating or touching the table with the peg, and re-insert it into the pegboard as quickly as possible, beginning with the top row and proceeding in a zigzag fashion through all 4 rows. One complete practice trial is performed to allow the child to learn the task, and the second trial is timed. The time taken to complete the test is measured with a stopwatch..

CONTACTS AND LOCATIONS:
Overall Officials: Emam EL-Negamy, PhD, Study Chair — Cairo University; Amira Mahmoud, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt